CLINICAL TRIAL: NCT02518100
Title: Vital Signs Patch: Early Feasibility and Usability Study - Feasibility Study for Automated Monitoring of Vital Signs Measurements in the In-Patient Hospital Setting
Brief Title: Vital Signs Patch: Automated Monitoring of Vital Signs Measurements in the In-Patient Hospital Setting
Acronym: VSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeWatch Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VSP-F004
Record Dates: First submitted 2015-08-03; First posted 2015-08-07 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Automated Measurement of Vital Signs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- VSP 3-Lead Study Participants (Experimental): Intervention: Vital Signs Patch (VSP) System 3-Lead (NEHB) Configuration The participants of this arm will have the following vital signs taken and recorded by the VSP System in the 3-lead (NEHB) configuration:
  Arterial blood oxygen Saturation (SpO2) ECG Heart Rate Surface Temperature Respiration
  Interventions: Device: Vital Signs Patch (VSP) System 3-Lead (NEHB) Configuration
- VSP 1-Lead Study Participants (Experimental): Intervention: Vital Signs Patch (VSP) System 1-Lead (PAL) Configuration. The participants of this arm will have the following vital signs taken and recorded by the VSP System in the 1-lead (PAL) configuration:
  Arterial blood oxygen Saturation (SpO2) ECG Heart Rate Surface Temperature Respiration
  Interventions: Device: Vital Signs Patch (VSP) System 1-Lead (PAL) Configuration

INTERVENTIONS:
Device: Vital Signs Patch (VSP) System 3-Lead (NEHB) Configuration — Vital signs will be taken using the Vital Signs Patch (VSP) System 3-Lead (NEHB) Configuration on each study participant in each Arm of this study for comparison against the same vital signs taken with traditional methods used by the facility.
  Arms: VSP 3-Lead Study Participants
Device: Vital Signs Patch (VSP) System 1-Lead (PAL) Configuration — Vital signs will be taken using the Vital Signs Patch (VSP) System 1-Lead (PAL) Configuration on each study participant in each Arm of this study for comparison against the same vital signs taken with traditional methods used by the facility.
  Arms: VSP 1-Lead Study Participants

SUMMARY:
This feasibility study evaluates the use of the Vital Signs Patch (VSP) System to take and monitor specified vital signs. It will be used in parallel with the normal equipment the study site uses to take and monitor vital signs.

DETAILED DESCRIPTION:
To assess the feasibility and usability of the total Vital Signs Patch (VSP) System in an actual hospital environment on in-patients by monitoring specified vital signs. The VSP System will be assessed for incorporation into the study site's Information Technology infrastructure. The VSP measurements will be compared with the predetermined expected results of the established vital signs equipment normally used by the facility based upon clinician protocols.

The VSP System can take and monitor patient vital signs in a more reliable and consistent manner by removing the human variability that occurs when clinicians manually take a patient's vital signs. The VSP has been designed to automatically take and monitor the following vital signs:

* Arterial blood oxygen Saturation (SpO2)
* ECG (up to 3 - Lead)
* Heart Rate (Part of ECG)
* Surface Temperature
* Respiration

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female hospital in-patients
* Vital signs considered 'stable' by clinical caregivers

Exclusion Criteria:

* Pediatric patients
* Female patients who are pregnant
* Patients with internal or external defibrillators
* Patients who have undergone surgery and still have a fresh incision on the chest
* Patients with skin damage on the chest such as burns, irritation, infections, wounds, etc.
* Patients who are in the Critical Care Unit (CCU)
* Patients who otherwise satisfy any of the contraindications associated with the VSP system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2016-08-16 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Composite Outcome Measure - Successful Vital Signs Acquisition | Up to Four Days
  Successful acquisition of Temperature, Heart Rate, ECG, Respiration, SpO2 daily for the inpatient stay of the subject up to four days. Success is achieved if all vital signs are obtained on a study participant. It is a composite result.

SECONDARY OUTCOMES:
Adhesion | Up to Four Days
  Successful performance of the adhesive of the vital signs patch during use on subjects. Adhesion will be measured as either positive or negative for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cantillon, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No